CLINICAL TRIAL: NCT00589355
Title: C-reactive Protein and Endothelial Dysfunction in Women With Glucose Intolerance
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Barbara I Gulanski, MD, MPH, Yale University School of Medicine
Other Study IDs: 12110
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Glucose Intolerance
Keywords: c-reactive protein; endothelial dysfunction; glucose intolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: postmenopausal women with glucose intolerance (either pre-diabetes or diet-controlled diabetes)
- 2: postmenopausal women with normal glucose tolerance

SUMMARY:
The goal of this study is to determine whether markers of vascular inflammation (such as c-reactive protein) can predict endothelial dysfunction (as measured by flow-mediated dilation) in postmenopausal women with glucose intolerance compared to normal controls.

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women
* ages 40-65

Exclusion Criteria:

* smokers
* diabetes requiring medication

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of healthy postmenopausal women who do not smoke. One group includes women with either pre-diabetes or diet-controlled diabetes. The control group includes women with normal glucose tolerance
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2002-01; Primary Completion 2003-06 (Actual); Study Completion 2008-10-01 (Actual)

PRIMARY OUTCOMES:
c-reactive protein | performed after screening evaluation

SECONDARY OUTCOMES:
flow-mediated dilation of brachial artery | performed twice after screening visit
sex steroids | performed after screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Gulanski, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States